CLINICAL TRIAL: NCT05623059
Title: Phase IIa Clinical Trial to Evaluate Pharmacokinetics and Safety of Slow Release DHEA
Brief Title: Evaluate Pharmacokinetics and Safety of Slow Release DHEA
Acronym: DHEA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kirsten Kloepfer, Associate Professor of Pediatrics, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15038; P01HL158507 (NIH)
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Asthma; Genotype
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This is an unblinded pharmacokinetic (PK) study to determine optimal dosing for future studies. This study will start with a one-time dose and progress to twice daily dosing for 3 days, every 12 hours. Study cohort will be 9 subjects with asthma. DHEA dose will be 50 mg via slow release capsules. Endpoints will be serum DHEA and DHEA-S levels at 10, 20, 30, 60 min & 2, 4, 6, 8, 12h after administration. After a one-week washout period, the protocol will be repeated using 100 mg of SR-DHEA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 50mg dose (Other): This arm will start with a one-time dose and progress to twice daily dosing for 3 days, every 12 hours. Study cohort will be 9 subjects with asthma. DHEA dose will be 50 mg via slow release capsules. Endpoints will be serum DHEA and DHEA-S levels at 10, 20, 30, 60 min & 2, 4, 6, 8, 12h after administration. After a one-week washout period, the protocol will be repeated using 100 mg of SR-DHEA.
  Interventions: Drug: Slow Release DHEA
- 100mg dose (Other): This arm will start with a one-time 100mg dose and progress to twice daily dosing for 3 days, every 12 hours. Study cohort will be same 9 subjects with asthma. DHEA dose will be 100mg via slow release capsules. Endpoints will be serum DHEA and DHEA-S levels at 10, 20, 30, 60 min & 2, 4, 6, 8, 12h after administration.
  Interventions: Drug: Slow Release DHEA

INTERVENTIONS:
Drug: Slow Release DHEA — DHEA is a hormone produced by the body's adrenal gland. In drug form, it is available as an over-the-counter supplement that is available on the market without prescription.
  Other Names: Slow Release Dehydroepiandrosterone

SUMMARY:
This is a study to look at pharmacokinetic levels of different doses of slow release DHEA in subjects with asthma.

DETAILED DESCRIPTION:
Pharmacokinetic (PK) studies of DHEA in asthma have never been done. In many diseases, PK in subjects with disease differs from that of control subjects and those with other conditions. Therefore, researchers are investigating if PK levels of slow release DHEA are different in subjects with asthma who have the HSD3B1 AA or AC phenotypes

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female aged between 18 and 50 at time of enrollment
* Evidence of asthma demonstrated by reversibility at visit 0 or by historical methacholine or bronchodilator reversibility if testing was performed under either the 2017 ERS technical standard (22) or the 1999 ATS Guidelines (23) or outside studies, provided that full sets of flow volume loops have been reviewed and approved by the PI. These criteria are defined as one of the following:
* For bronchodilator reversibility: An increase in FEV1 ≥10% (24) compared to the baseline (and 200 ml) after up to 8 puffs of albuterol
* For historical methacholine responsiveness: Positive methacholine defined as PC20 ≤ 16 mg/ml, or PD20 ≤400 mcg
* Physician diagnosis of asthma according to NHLBI guidelines;
* Consistent use of an ICS/LABA inhaler for the prior 2 months;
* Non smoker;
* Females must not be pregnant or lactating;
* Absence of non-allergic comorbidities;
* Genotype testing positive for either HSD3B1 AA or AC specific variant

Exclusion Criteria:

* Pregnant or actively trying to become pregnant; breastfeeding
* positive urine pregnancy test
* Known lung disease other than asthma
* Acute (non asthma-related) dyspnea, viral respiratory illness or asthma exacerbation within 4 weeks of screening
* Systemic glucocorticoid dosing for maintenance >10 mg/day of prednisone or equivalent
* Patients with significant non-allergic comorbidities (e.g. cerebral palsy, heart disease, kidney disease, liver disease, etc.)
* Patients with any know central or peripheral endocrine abnormality such as precocious puberty or diabetes
* Patients with any known previous adverse reaction to DHEA
* Current smoker or pack year history > 5 years (includes vaping/nicotine inhalation devices)
* Positive urine cotinine test (> 100 mg/mL)
* Use of prednisone or antibiotics in the last 4 weeks
* Use of any performance-enhancing drugs in the last 2 weeks
* Use of DHEA in the last 2 weeks
* Androgen use for any reason
* HSD3B1 CC phenotype
* Any other condition or finding that would compromise the safety of the subject or the quality of the study data, or otherwise interfere with achieving the study objectives, as determined by the PI
* Menopausal amenorrhea by history
* Positive PSA (>4 ng/ml) (Prostate Specific Antigen)
* Prior diagnosis of vocal cord dysfunction, bronchopulmonary dysplasia, cystic fibrosis, chronic obstructive pulmonary disorder, or other lung disease
* Systolic blood pressure > 150 mm Hg and/or diastolic blood pressure >90 mm Hg
* Heart rates outside the range of 50 to 120 beats per minutes or with a pathologic irregularity
* Patients afflicted with any additional acute or chronic pathology that in the opinion of the screening physician makes them unsuitable for study or increases the risks associated with the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose for slow release DHEA in asthmatic subjects on a single and recurring regimen of 50mg and of 100mg by pharmacokinetic evaluation. | From baseline to 12 hours after the final dose (up to 66 days)
  The objective is to determine the maximum tolerated dose of slow release DHEA in patients with asthma and AA or AC genotype by measuring the presence in and difference of pharmacokinetics of two dose levels (50mg and 100mg).
Determine the maximum tolerated dose for slow release DHEA for asthmatic subjects on a regimen of 50mg and 100mg by adverse event evaluation. | From administration of the first dose to 12 hours after the final dose (up to 59 days)]
  The objective is to determine the maximum tolerated dose of slow release DHEA in patients with asthma and AA or AC genotype by evaluating the occurrences and severity of adverse events during or after dosing at two levels (5omg and 100mg).

SECONDARY OUTCOMES:
Safety and tolerability evaluation measured by the change in vital signs from baseline to post-treatment (Vital signs will include heart-rate, respiratory rate, RA saturation) | From baseline to after the first washout period (up to 63 days)]
  The objective is to evaluate the safety and tolerability of slow release DHEA in asthma by measuring the change in vital signs from before treatment to after treatment.
Safety and tolerability evaluation measured by a change in physical symptoms from baseline to post-treatment. Physical symptoms will include reports such as cough, shortness of breath, chest tightness, wheeze) | From baseline to after the first washout period (up to 63 days)]
  The objective is to evaluate the safety and tolerability of slow release DHEA in asthma by measuring the change in physical symptoms from before treatment to after treatment.
Safety and tolerability evaluation measured by the change in physical exam findings from baseline to post-treatment | From baseline to after the first washout period (up to 63 days)
  The objective is to evaluate the safety and tolerability of slow release DHEA in asthma by measuring the change in physical exam findings from before treatment to after treatment.
Safety and tolerability evaluation measured by the change in FEV from baseline to post-treatment (as measured by spirometry). | From baseline to after the first washout period (up to 63 days)
  The objective is to evaluate the safety and tolerability of slow release DHEA in asthma patients by performing pulmonary function testing to obtain measurements of FEV (forced expiratory volume) before treatment and after treatment.
Safety and tolerability evaluation measured by the occurrence of an asthma exacerbation event during and after treatment. | From administration of the first dose to 12 hours after the final dose (up to 59 days)
  The objective is to evaluate the safety and tolerability of slow release DHEA in asthma patients by recording any instance of asthma exacerbation event during or after treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Riley Hospital for Children, Indianapolis, Indiana
  - University Hospital, Indianapolis, Indiana

REFERENCES:
- [Background] Sadatsafavi M, Lynd L, Marra C, Carleton B, Tan WC, Sullivan S, Fitzgerald JM. Direct health care costs associated with asthma in British Columbia. Can Respir J. 2010 Mar-Apr;17(2):74-80. doi: 10.1155/2010/361071. PMID 20422063
- [Background] Han MK, Arteaga-Solis E, Blenis J, Bourjeily G, Clegg DJ, DeMeo D, Duffy J, Gaston B, Heller NM, Hemnes A, Henske EP, Jain R, Lahm T, Lancaster LH, Lee J, Legato MJ, McKee S, Mehra R, Morris A, Prakash YS, Stampfli MR, Gopal-Srivastava R, Laposky AD, Punturieri A, Reineck L, Tigno X, Clayton J. Female Sex and Gender in Lung/Sleep Health and Disease. Increased Understanding of Basic Biological, Pathophysiological, and Behavioral Mechanisms Leading to Better Health for Female Patients with Lung Disease. Am J Respir Crit Care Med. 2018 Oct 1;198(7):850-858. doi: 10.1164/rccm.201801-0168WS. PMID 29746147
- [Background] Zein JG, Erzurum SC. Asthma is Different in Women. Curr Allergy Asthma Rep. 2015 Jun;15(6):28. doi: 10.1007/s11882-015-0528-y. PMID 26141573
- [Background] Zein J, Gaston B, Bazeley P, DeBoer MD, Igo RP Jr, Bleecker ER, Meyers D, Comhair S, Marozkina NV, Cotton C, Patel M, Alyamani M, Xu W, Busse WW, Calhoun WJ, Ortega V, Hawkins GA, Castro M, Chung KF, Fahy JV, Fitzpatrick AM, Israel E, Jarjour NN, Levy B, Mauger DT, Moore WC, Noel P, Peters SP, Teague WG, Wenzel SE, Erzurum SC, Sharifi N. HSD3B1 genotype identifies glucocorticoid responsiveness in severe asthma. Proc Natl Acad Sci U S A. 2020 Jan 28;117(4):2187-2193. doi: 10.1073/pnas.1918819117. Epub 2020 Jan 13. PMID 31932420
- [Background] Marozkina N, Zein J, DeBoer MD, Logan L, Veri L, Ross K, Gaston B. Dehydroepiandrosterone Supplementation May Benefit Women with Asthma Who Have Low Androgen Levels: A Pilot Study. Pulm Ther. 2019 Dec;5(2):213-220. doi: 10.1007/s41030-019-00101-9. Epub 2019 Oct 21. PMID 32026412
- [Background] Lahm T, Albrecht M, Fisher AJ, Selej M, Patel NG, Brown JA, Justice MJ, Brown MB, Van Demark M, Trulock KM, Dieudonne D, Reddy JG, Presson RG, Petrache I. 17beta-Estradiol attenuates hypoxic pulmonary hypertension via estrogen receptor-mediated effects. Am J Respir Crit Care Med. 2012 May 1;185(9):965-80. doi: 10.1164/rccm.201107-1293OC. Epub 2012 Mar 1. PMID 22383500
- [Background] Bentley JK, Hershenson MB. Airway smooth muscle growth in asthma: proliferation, hypertrophy, and migration. Proc Am Thorac Soc. 2008 Jan 1;5(1):89-96. doi: 10.1513/pats.200705-063VS. PMID 18094090
- [Background] Chang KH, Li R, Kuri B, Lotan Y, Roehrborn CG, Liu J, Vessella R, Nelson PS, Kapur P, Guo X, Mirzaei H, Auchus RJ, Sharifi N. A gain-of-function mutation in DHT synthesis in castration-resistant prostate cancer. Cell. 2013 Aug 29;154(5):1074-1084. doi: 10.1016/j.cell.2013.07.029. PMID 23993097
- [Background] Hall SL, Baker T, Lajoie S, Richgels PK, Yang Y, McAlees JW, van Lier A, Wills-Karp M, Sivaprasad U, Acciani TH, LeCras TD, Myers JB, Kovacic MB, Lewkowich IP. IL-17A enhances IL-13 activity by enhancing IL-13-induced signal transducer and activator of transcription 6 activation. J Allergy Clin Immunol. 2017 Feb;139(2):462-471.e14. doi: 10.1016/j.jaci.2016.04.037. Epub 2016 Jun 11. PMID 27417023
- [Background] Bulitta JB, Jiao Y, Drescher SK, Oliver A, Louie A, Moya B, Tao X, Wittau M, Tsuji BT, Zavascki AP, Shin BS, Drusano GL, Sorgel F, Landersdorfer CB. Four Decades of beta-Lactam Antibiotic Pharmacokinetics in Cystic Fibrosis. Clin Pharmacokinet. 2019 Feb;58(2):143-156. doi: 10.1007/s40262-018-0678-x. PMID 29936678
- [Background] Hettel D, Zhang A, Alyamani M, Berk M, Sharifi N. AR Signaling in Prostate Cancer Regulates a Feed-Forward Mechanism of Androgen Synthesis by Way of HSD3B1 Upregulation. Endocrinology. 2018 Aug 1;159(8):2884-2890. doi: 10.1210/en.2018-00283. PMID 29850791
- [Background] Gaston B, Reilly J, Drazen JM, Fackler J, Ramdev P, Arnelle D, Mullins ME, Sugarbaker DJ, Chee C, Singel DJ, Loscalzo J, Stamler JS. Endogenous nitrogen oxides and bronchodilator S-nitrosothiols in human airways. Proc Natl Acad Sci U S A. 1993 Dec 1;90(23):10957-61. doi: 10.1073/pnas.90.23.10957. PMID 8248198
- [Background] Gaston B, Sears S, Woods J, Hunt J, Ponaman M, McMahon T, Stamler JS. Bronchodilator S-nitrosothiol deficiency in asthmatic respiratory failure. Lancet. 1998 May 2;351(9112):1317-9. doi: 10.1016/S0140-6736(97)07485-0. PMID 9643794
- [Background] Hunt JF, Fang K, Malik R, Snyder A, Malhotra N, Platts-Mills TA, Gaston B. Endogenous airway acidification. Implications for asthma pathophysiology. Am J Respir Crit Care Med. 2000 Mar;161(3 Pt 1):694-9. doi: 10.1164/ajrccm.161.3.9911005. PMID 10712309
- [Background] Carraro S, Doherty J, Zaman K, Gainov I, Turner R, Vaughan J, Hunt JF, Marquez J, Gaston B. S-nitrosothiols regulate cell-surface pH buffering by airway epithelial cells during the human immune response to rhinovirus. Am J Physiol Lung Cell Mol Physiol. 2006 May;290(5):L827-32. doi: 10.1152/ajplung.00406.2005. PMID 16603595
- [Background] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Background] Watson AC, Rosenfield RL, Fang VS. Recovery from glucocorticoid inhibition of the responses to corticotrophin-releasing hormone. Clin Endocrinol (Oxf). 1988 May;28(5):471-7. doi: 10.1111/j.1365-2265.1988.tb03681.x. PMID 2850875
- [Background] Jollin L, Thomasson R, Le Panse B, Baillot A, Vibarel-Rebot N, Lecoq AM, Amiot V, De Ceaurriz J, Collomp K. Saliva DHEA and cortisol responses following short-term corticosteroid intake. Eur J Clin Invest. 2010 Feb;40(2):183-6. doi: 10.1111/j.1365-2362.2009.02219.x. Epub 2009 Oct 29. PMID 19874391
- [Background] Al-Tarrah K, Moiemen N, Lord JM. The influence of sex steroid hormones on the response to trauma and burn injury. Burns Trauma. 2017 Sep 14;5:29. doi: 10.1186/s41038-017-0093-9. eCollection 2017. PMID 28920065
- [Background] Phipatanakul W, Mauger DT, Sorkness RL, Gaffin JM, Holguin F, Woodruff PG, Ly NP, Bacharier LB, Bhakta NR, Moore WC, Bleecker ER, Hastie AT, Meyers DA, Castro M, Fahy JV, Fitzpatrick AM, Gaston BM, Jarjour NN, Levy BD, Peters SP, Teague WG, Fajt M, Wenzel SE, Erzurum SC, Israel E; Severe Asthma Research Program. Effects of Age and Disease Severity on Systemic Corticosteroid Responses in Asthma. Am J Respir Crit Care Med. 2017 Jun 1;195(11):1439-1448. doi: 10.1164/rccm.201607-1453OC. PMID 27967215
- [Background] Coates AL, Wanger J, Cockcroft DW, Culver BH; Bronchoprovocation Testing Task Force: Kai-Hakon Carlsen; Diamant Z, Gauvreau G, Hall GL, Hallstrand TS, Horvath I, de Jongh FHC, Joos G, Kaminsky DA, Laube BL, Leuppi JD, Sterk PJ. ERS technical standard on bronchial challenge testing: general considerations and performance of methacholine challenge tests. Eur Respir J. 2017 May 1;49(5):1601526. doi: 10.1183/13993003.01526-2016. Print 2017 May. PMID 28461290
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999 Jan;159(1):179-87. doi: 10.1164/ajrccm.159.1.9712108. PMID 9872837
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880

DOCUMENTS (1):
  • Informed Consent Form (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT05623059/ICF_000.pdf